CLINICAL TRIAL: NCT02760901
Title: Evaluation of the Effect of Acetazolamide, Mannitol and N-acetylcysteine on Cisplatin-Induced Nephrotoxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Kamal Morsy Ibraheem, clinical pharmacist, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: master
Record Dates: First submitted 2016-04-01; First posted 2016-05-04 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Cisplatin Nephrotoxicity
MeSH Terms: interventions — Acetazolamide; Acetylcysteine; Mannitol; Sodium Chloride; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mannitol group (Active Comparator): patients received mannitol 20 % 100 ml half an hour before cisplatin and saline hydration.
  Interventions: Drug: Mannitol; Drug: saline; Drug: Cisplatin
- ACTZ group (Active Comparator): patients received acetazolamide 250 mg half an hour before cisplatin with saline hydration.
  Interventions: Drug: Acetazolamide; Drug: saline; Drug: Cisplatin
- NAC group (Active Comparator): patients received acetylcysteine NAC (600 mg every 12 hours) for 4 doses beginning 24 hours before cisplatin with saline hydration.
  Interventions: Drug: Acetylcysteine; Drug: saline; Drug: Cisplatin

INTERVENTIONS:
Drug: Acetazolamide — patients received acetazolamide 250 mg half an hour before cisplatin with saline hydration.for prevention of cisplatin nephrotoxicity
  Other Names: ACTZ
  Arms: ACTZ group
Drug: Acetylcysteine — patients received NAC (600 mg every 12 hours) for 4 doses beginning 24 hours before cisplatin with saline hydration.for prevention of cisplatin nephrotoxicity
  Other Names: NAC
  Arms: NAC group
Drug: Mannitol — patients received mannitol 20 % 100 ml half an hour before cisplatin and saline hydration.
  Arms: Mannitol group
Drug: saline — saline hydration 2500 ml before cisplatin therapy
Drug: Cisplatin — patients with tumours already prescribed cisplatin

SUMMARY:
Cisplatin is a major anti-neoplastic drug used for the treatment of solid tumors. Its chief dose limiting side effect is nephrotoxicity. Twenty percent of patients receiving high-dose cisplatin undergo severe renal dysfunction. Acetazolamide and N-acetylcysteine (NAC) ameliorated Cisplatin-induced nephrotoxicity in rats. No study to date evaluated the protective effect of acetazolamide or NAC against cisplatin nephrotoxicity in humans.

Aim of the study was to evaluate the effect of acetazolamide or NAC against cisplatin nephrotoxicity in humans compared to mannitol and to each other.

Patients and methods. A total 52 patients receiving standard hydration measures for cisplatin were randomized to three groups: 20 patients receiving mannitol, 15 patients receiving acetazolamide and 17 patients receiving NAC. Patients' kidney function was monitored using serum creatinine, creatinine clearance and blood urea nitrogen; kidney injury was assessed using RIFLE criteria. Patients' liver function tests and hematological parameters were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients to receive cisplatin based chemotherapy protocol.
2. Adult patients from 18 to 65 years.

Exclusion Criteria:

1. Existing renal impairment ( Creatinine clearance <30 ml/minute)
2. Severe hepatic impairment (Child Pugh score C).
3. Hypersensitivity to sulfonamides.
4. Patients with chronic non-congestive angle closure glaucoma.
5. Hypersensitivity to sulphur compounds, N-acetylcysteine or any component of the formulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Serum Creatinine | change from baseline after 3 cycles separated by 21 days
  Blood samples collected and measured in laboratory with the unit mg/dL
Creatinine clearance according to Cockroft-Gault equation | change from baseline after 3 cycles separated by 21 days
  calculated using globalrph calculators , unit ml/min
Acute kidney injury | change from baseline after 3 cycles separated by 21 days
  Acute kidney injury assessed by RIFLE criteria that was calculated for patients
Blood urea nitrogen (BUN) | change from baseline after 3 cycles separated by 21 days
  Blood samples collected and measured in laboratory with the unit mg/dl

SECONDARY OUTCOMES:
Aspartate Transaminase (AST) | change from baseline after 3 cycles separated by 21 days
  Liver function tests were monitored by measuring AST for change from baseline after 3 cycles separated by 21 days
hemoglo bin | change from baseline after 3 cycles separated by 21 days
  hemoglobin concentration g/dl was monitored for change from baseline after 3 cycles separated by 21 days
adverse events | change from baseline after 3 cycles separated by 21 days
  Monitoring adverse events: to evaluate the difference between three groups regarding frequency of adverse events.
Alanine Transaminase (ALT) | change from baseline after 3 cycles separated by 21 days
  Liver function tests were monitored by measuring ALT for change from baseline after 3 cycles separated by 21 days
platelets count | change from baseline after 3 cycles separated by 21 days
  platelets count cells per ml was monitored for change from baseline after 3 cycles separated by 21 days
total leucocyte count | change from baseline after 3 cycles separated by 21 days
  total leucocyte count cells per ml was monitored for change from baseline after 3 cycles separated by 21 days